CLINICAL TRIAL: NCT07270107
Title: Immersive Virtual Reality Versus Traditional Instruction for Teaching the Bobath Concept in Physiotherapy Education: A Randomized Controlled Trial
Brief Title: Bobath Instruction in Physiotherapy: Virtual Reality Versus Traditional Methods
Acronym: BOBATH-PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Sağlık ve Teknoloji Üniversitesi (Other)
Responsible Party: Principal Investigator, Sena Çınarlı, Asisstant Professor, Kocaeli Sağlık ve Teknoloji Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KOSTU-25-BOBATH
Record Dates: First submitted 2025-11-22; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Physical Therapy; Education; Virtual Reality; Neurorehabilitation
Keywords: Neurorehabilitation; Immersive virtual reality; Objective Structured Clinical Examination; Digital health education

STUDY DESIGN:
Intervention Model Description: This study used a two-arm, parallel-group, single-blind randomized controlled trial design comparing immersive virtual reality-based instruction with traditional face-to-face education for teaching the Bobath concept to physiotherapy students. Participants were randomly allocated in a 1:1 ratio, and blinded evaluators conducted all theoretical and practical assessments at post-test and retention time points.
Who Masked: Outcomes Assessor
Masking Description: This study used a single-blind design in which outcome assessors were blinded to group allocation. Participants, care providers, and investigators were not blinded due to the nature of the educational intervention."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-Face Bobath Instruction (Active Comparator): Participants assigned to the Face-to-Face (F2F) group received a 45-minute instructor-led session consisting of theoretical explanation and practical demonstrations of Bobath-based postural control strategies. The session included live demonstration of facilitation techniques, alignment correction, and trunk control activities. After the instructional segment, students practiced the techniques in small groups under instructor supervision. Content duration, learning objectives, and practice structure were standardized across both study arms.
  Interventions: Other: Traditional instruction
- Virtual Reality Bobath Instruction (Experimental): Participants in the Virtual Reality (VR) group received the same 45-minute instructional content through an immersive 360° VR video recorded by the same instructor. The VR session integrated theoretical narration with practical demonstrations of Bobath postural control strategies. Students viewed the session collectively using VR headsets. A structured debriefing followed to reinforce key concepts and allow question clarification. As in the F2F group, students then practiced the techniques in small groups following the session.
  Interventions: Device: Immersive VR headset instruction

INTERVENTIONS:
Device: Immersive VR headset instruction — The study interventions consisted of two educational delivery methods used to teach the Bobath concept in physiotherapy training. Both interventions provided identical learning objectives, theoretical content, and practical demonstration elements related to postural control strategies. The instructional materials were standardized in duration, sequencing, and educational objectives to ensure equivalence across groups. Delivery differed only in format, with one method provided through traditional in-person instruction and the other through immersive virtual reality technology. All students practiced the demonstrated techniques following the instructional component, and no additional instructional materials were provided beyond the assigned modality
  Arms: Virtual Reality Bobath Instruction
Other: Traditional instruction — This intervention delivers Bobath concept education through conventional face-to-face teaching methods. The instructional session includes faculty-led theoretical explanations and live demonstrations delivered in a traditional classroom or laboratory setting. Students receive the standardized content through direct instructor interaction, consistent with customary physiotherapy training practices. All participants subsequently engage in supervised practice to apply the demonstrated concepts.
  Arms: Face-to-Face Bobath Instruction

SUMMARY:
This randomized controlled trial evaluated the effectiveness of immersive virtual reality (VR)-based instruction compared with traditional face-to-face teaching for delivering the Bobath concept in physiotherapy education. Third-year physiotherapy students were randomly assigned to either VR-based or conventional instruction and completed standardized theoretical and practical assessments immediately after training and again two weeks later. While both instructional methods resulted in comparable short-term learning outcomes, the VR group demonstrated superior retention of practical skills at follow-up. Findings suggest that immersive VR is a feasible and effective educational approach for enhancing motor skill learning in neurophysiological rehabilitation training.

DETAILED DESCRIPTION:
This two-arm, parallel-group, single-blind randomized controlled trial aims to investigate whether immersive virtual reality (VR)-based education can enhance learning and retention of the Bobath concept among undergraduate physiotherapy students. The Bobath approach, widely used in neurorehabilitation, requires learners to integrate postural control principles, movement facilitation techniques, and sensorimotor strategies-skills traditionally taught through face-to-face lectures and hands-on demonstrations. Given the increasing integration of digital technologies in health professions education, immersive VR may offer an alternative through interactive, high-fidelity, and repeatable learning experiences.

Students will be randomized to receive either a standardized face-to-face instructional session or an immersive 360° VR-based session of equivalent duration and content. Both groups will be exposed to theoretical explanations and practical demonstrations focusing on trunk control strategies, alignment principles, and facilitation techniques. Practical components in both groups will be reinforced through structured small-group practice following the instructional session.

To ensure methodological rigor, two independent evaluators blinded to group allocation will assess student performance through a multiple-choice knowledge test and a three-station Objective Structured Clinical Examination (OSCE), administered two days after training and again two weeks later to evaluate retention. Inter-rater reliability will be calculated to ensure consistency of scoring across evaluators.

ELIGIBILITY:
Inclusion Criteria:

* Third-year undergraduate physiotherapy students.
* First-time enrollment in the Neurophysiological Approaches II course.
* No prior training or formal exposure to the Bobath concept.
* System Usability Scale (SUS) score classified as A+ (96-100 percentile). -Ability to participate in VR or face-to-face instruction as assigned.- Voluntary participation with provision of written informed consent.-

Exclusion Criteria:

* History of medical conditions contraindicating VR use (e.g., vestibular disorders, migraine, epilepsy).
* Prior experience, certification, or coursework related to the Bobath concept.
* Failure to provide informed consent.
* Any condition that may limit safe participation in the educational session or assessments.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Theoretical Knowledge Score | Post-test at 2 days and retention test at 2 weeks after the intervention
  Description:
  The theoretical outcome measure assesses students' understanding of Bobath-based postural control strategies using a 10-item multiple-choice examination. Each correct response is awarded 1 point. Raw scores (0-10) are converted to a 0-100 scale.
  Score Range: 0-100 Direction: Higher scores indicate better theoretical knowledge. The same standardized test is administered at both assessment points to evaluate learning and retention under the two instructional modalities.
Practical Performance Score (OSCE) | Post-test at 2 days and retention test at 2 weeks after the intervention
  Practical skill performance is evaluated using a three-station Objective Structured Clinical Examination (OSCE) assessing Bobath-based postural control strategies. Each station uses a standardized 3-point checklist (0 = not performed, 1 = partially performed, 2 = correctly performed). The combined station scores are converted to a 0-100 scale.
  Score Range: 0-100 Direction: Higher scores indicate better practical performance. All assessments are video-recorded and independently scored by two blinded evaluators using the same scoring rubric. This metric evaluates both immediate skill acquisition and subsequent retention.

OTHER OUTCOMES:
Inter-Rater Reliability of Practical Performance Scores | At post-test (2 days) and retention (2 weeks)
  Inter-rater reliability of OSCE practical performance scores is assessed using the Intraclass Correlation Coefficient (ICC, two-way random effects, absolute agreement) and Cohen's kappa for pass/fail classification. These metrics evaluate the consistency and agreement between the two blinded evaluators scoring the practical examinations.
Pass/Fail Classification Based on Combined Score | Post-test at 2 days and retention test at 2 weeks
  Students' overall performance is classified as pass or fail based on a predefined threshold of ≥70% from combined theoretical and practical scores. Pass rates are compared between groups to assess competency achievement in each instructional modality.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Sena Çınarlı, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli Health and Technology University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not yet determined whether individual participant data (IPD) will be shared. A decision regarding data sharing will be made after study completion, considering institutional policies, ethical requirements, and data privacy standards.